CLINICAL TRIAL: NCT04889274
Title: A Double-blind, Randomised, Placebo-controlled Parallel Study to Investigate the Effect of Dietary Nitrate and Sex on COVID-19 Vaccine Induced Vascular Dysfunction in Healthy Men and Women
Brief Title: Investigation of the Effects of Dietary Nitrate and Sex on COVID-19 Vaccine Induced Vascular Dysfunction in Healthy Men and Women (DiNOVasc-COVID-19)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 21/SC/0154
Record Dates: First submitted 2021-05-06; First posted 2021-05-17 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular Diseases; Endothelial Dysfunction
Keywords: COVID-19, endothelial dysfunction, nitrate, nitrite, sex
MeSH Terms: conditions — Cardiovascular Diseases; COVID-19; Coitus | interventions — COVID-19 Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A: Male healthy volunteers (Experimental)
  Interventions: Biological: COVID-19 vaccine
- Part A: Female healthy volunteers (Experimental)
  Interventions: Biological: COVID-19 vaccine
- Part B: Nitrate-rich beetroot juice (Active Comparator): Dietary Supplement: Concentrate beetroot Juice (70 ml) containing ~5mmol of inorganic nitrate
  Interventions: Biological: COVID-19 vaccine; Biological: Concentrate beetroot Juice
- Part B: Nitrate-deplete beetroot juice (Placebo Comparator): Dietary Supplement: Concentrate beetroot Juice (70 ml) which is nitrate-depleted
  Interventions: Biological: COVID-19 vaccine; Biological: Nitrate-deplete beetroot juice

INTERVENTIONS:
Biological: COVID-19 vaccine — COVID-19 vaccine as offered by NHS England
Biological: Concentrate beetroot Juice — Beetroot juice containing approximately 5mmol/l nitrate
  Arms: Part B: Nitrate-rich beetroot juice
Biological: Nitrate-deplete beetroot juice — Beetroot juice with nitrate removed
  Arms: Part B: Nitrate-deplete beetroot juice

SUMMARY:
Inorganic nitrate can protect blood vessels from the damage that occurs during cardiovascular disease. Early experimental work suggests that nitrate-induced improvements in vascular function relate to the suppression of inflammatory pathways. Whether this protection against inflammation-induced damage to the blood vessel wall might also be functional in the setting of COVID-19 vaccination will be investigated.

Vascular function will be assessed before and after the healthy participant has received their COVID-19-vaccination. Whether there might be differences in the response to the vaccine between the sexes and whether a dietary nitrate intervention impacts upon the effects of vaccination will be investigated.

The study is in two parts:

Part A: To assess sex differences in the vascular response to COVID-19 vaccination.

Part B: To assess whether inorganic nitrate, in the form of dietary inorganic nitrate supplementation compared to placebo control, can raise circulating plasma nitrite levels and thereby prevent the systemic inflammation that causes vascular dysfunction.

DETAILED DESCRIPTION:
Whether the COVID-19 vaccine can be used to study endothelial dysfunction and whether inorganic nitrate might be useful in restoring the function of the endothelium in a scenario simulating the COVID-19 infection setting will be investigated.

Furthermore, sex differences in the vascular response to the COVID-19 vaccination will be investigated.

Design: A prospective randomised, double-blind, placebo-controlled trial.

Target population: A total of 98 healthy participants will be recruited. Part A: 30 participants (15 male, 15 female.) Part B: 68 participants (34 intervention, 34 placebo). Participants will be recruited prior to receiving the COVID-19 vaccination, via Barts Health NHS Trust approved vaccination hubs.

Setting: Equal numbers of healthy male and female volunteers, aged between 18 and 60 years of age, will be recruited. Following recruitment, participants will undergo baseline measurements of vascular function of flow mediated dilatation (FMD) and pulse wave analysis/velocity (PWA, PWV), in addition to haematological and clinical biochemical analyses. Volunteers will then be randomised into one of the 2 study Parts (Part A: sex differences in vascular response to COVID-19 vaccine, Part B: influence of dietary nitrate upon vascular responses to COVID-19 vaccine). If randomised to Part B, volunteers will be treated with 3 days of either 4-5mmol nitrate-containing beetroot juice or placebo. If randomised to Part A, the volunteers will not receive an intervention. On day 3, all participants will receive their COVID-19 vaccine. At 8±2hours after the vaccine, the participants will undergo repeat measurements of vascular function. A quality of life questionnaire will be obtained 28 days after the vaccine has been administered.

Intervention: All volunteers will receive COVID-19 vaccination in Part A and Part B. In Part B of the study, volunteers will be randomised in a 1:1 fashion to receive either nitrate-containing beetroot juice (4-5mmol nitrate) or nitrate-deplete placebo.

The study will take place in the Clinical Research Centre at The William Harvey Research Institute.

Analysis: For the analysis of Part A linear regression will be used to compare change in vascular dysfunction from pre- to post-vaccination between the sexes, unadjusted and adjusted for important risk factors including age, BMI and baseline vessel diameter. For Part B analysis of covariance (ANCOVA) will be used to compare change in vascular dysfunction from pre- to post-vaccination between dietary nitrate and placebo control groups adjusting for pre-vaccination level, and to compare change in plasma nitrite between dietary nitrate and placebo control groups adjusting for baseline nitrite level.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers with a booking for COVID-19 vaccination slot as per government guidelines
2. Aged 18-60
3. Volunteers who are willing to sign the consent form

Exclusion Criteria:

1. Aged <18 or >60 years
2. Healthy subjects unwilling to consent
3. Pregnant, or any possibility that a subject may be pregnant
4. History of any serious illnesses, including recent infections or trauma
5. Subjects taking systemic medication (other than the oral contraceptive pill)
6. Subjects with self-reported use of mouthwash or tongue scrapes
7. Subjects with recent (2 weeks) or current antibiotic use
8. Subjects with a history, or recent treatment of (within last 3 months) any oral condition (excluding caries), including gingivitis, periodontitis and halitosis
9. Subjects with a history of COVID-19 vaccination
10. Subjects with any history of a blood-borne infectious

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of change in FMD from baseline between the sexes after COVID-19 vaccination | Up to 28 days
  A measurement of brachial artery diameter using ultrasound (FMD, flow mediated dilatation) will be conducted at visits 2 and 3 (i.e. pre- and post-vaccine). This outcome measure will compare these 2 measurements, and change in FMD will be calculated as subtracting the value collected at visit 3 from visit 2, and expressed as a percentage (%). Comparisons will then be made between the sexes (i.e. males vs females) in Part A.
Comparison of change in FMD from baseline after COVID-19 vaccination following inorganic nitrate versus placebo supplementation | Up to 28 days
  A measurement of brachial artery diameter using ultrasound (FMD, flow mediated dilatation) will be conducted at visits 2 and 3 (i.e. pre- and post-vaccine). This outcome measure will compare these 2 measurements, and change in FMD will be calculated as subtracting the value collected at visit 3 from visit 2, and expressed as a percentage (%). Comparisons will then be made between intervention and placebo in Part B.
Comparison of change in plasma [NO2-] following inorganic nitrate versus placebo supplementation | Up to 28 days
  Quantification of [NO2-] will be made using ozone chemiluminescence. Samples of blood, urine and saliva will be acquired at visit 2 and visit 3 (i.e. pre- and post-vaccine). Measurement of [NO2-] will be made in all matrices at both timepoints, and a comparison will be made (for this we plan on using 2-way ANOVA, using GraphPad Prism statistics package) to compare time and intervention.

SECONDARY OUTCOMES:
Comparison between the sexes in the systemic inflammatory response to COVID-19 vaccination | Up to 28 days
  Comparisons of the inflammatory response will be made using a combination of clinical haematology and chemistry to assess leukocyte sub-types, and inflammatory markers such as C-reactive protein. Samples of blood will be acquired at visit 2 and visit 3 (i.e. pre- and post-vaccine). Comparison will be made (for this we plan on using 2-way ANOVA, using GraphPad Prism statistics package) to compare time and intervention.
Comparison between nitrate and placebo with respect to inflammatory cell activation state | Up to 28 days
  Comparisons of the inflammatory cell activation state will be made through the assessment of inflammatory cytokines and chemokines (bead array analyser). Samples of blood plasma will be acquired at visit 2 and visit 3 (i.e. pre- and post-vaccine). Comparison will be made (for this we plan on using 2-way ANOVA, using GraphPad Prism statistics package) to compare time and intervention.
Comparison between nitrate and placebo with respect to circulating inflammatory mediators | Up to 28 days
  Comparisons of the inflammatory mediators will be made through the assessment of inflammatory cytokines and chemokines (bead array analyser). Samples of blood plasma will be acquired at visit 2 and visit 3 (i.e. pre- and post-vaccine). Comparison will be made (for this we plan on using 2-way ANOVA, using GraphPad Prism statistics package) to compare time and intervention.
Comparison between nitrate and placebo with respect to platelet function during systemic inflammation | Up to 28 days
  Comparisons of the platelet function will be made through the use of a platelet aggregometer and flow cytometry. Samples of citrate containing whole blood will be acquired at visit 2 and visit 3 (i.e. pre- and post-vaccine). Comparison will be made (for this we plan on using 2-way ANOVA, using GraphPad Prism statistics package) to compare time and intervention.
Comparison between nitrate and placebo with respect to endothelium independent vasodilation of the brachial artery | Up to 28 days
  Comparisons of endothelium independent vascular function will be made through the use brachial artery ultrasound and sublingual glyceryl trinitrate. Vascular ultrasound will be conducted at visit 2 and visit 3 (i.e. pre- and post-vaccine). Comparison will be made (for this we plan on using 2-way ANOVA, using GraphPad Prism statistics package) to compare time and intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- The William Harvey Research Institute, London, United Kingdom

REFERENCES:
- [Result] Rathod KS, Kapil V, Velmurugan S, Khambata RS, Siddique U, Khan S, Van Eijl S, Gee LC, Bansal J, Pitrola K, Shaw C, D'Acquisto F, Colas RA, Marelli-Berg F, Dalli J, Ahluwalia A. Accelerated resolution of inflammation underlies sex differences in inflammatory responses in humans. J Clin Invest. 2017 Jan 3;127(1):169-182. doi: 10.1172/JCI89429. Epub 2016 Nov 28. PMID 27893465
- [Result] Kapil V, Khambata RS, Jones DA, Rathod K, Primus C, Massimo G, Fukuto JM, Ahluwalia A. The Noncanonical Pathway for In Vivo Nitric Oxide Generation: The Nitrate-Nitrite-Nitric Oxide Pathway. Pharmacol Rev. 2020 Jul;72(3):692-766. doi: 10.1124/pr.120.019240. PMID 32576603
- [Result] Shabbir A, Rathod KS, Khambata RS, Ahluwalia A. Sex Differences in the Inflammatory Response: Pharmacological Opportunities for Therapeutics for Coronary Artery Disease. Annu Rev Pharmacol Toxicol. 2021 Jan 6;61:333-359. doi: 10.1146/annurev-pharmtox-010919-023229. Epub 2020 Oct 9. PMID 33035428
- [Derived] Shabbir A, Chhetri I, Khambata RS, Parakaw T, Lau C, Aubdool MABN, Massimo G, Dyson N, Kapil V, Godec T, Apea V, Flint J, Orkin C, Rathod KS, Ahluwalia A. A double-blind, randomised, placebo-controlled parallel study to investigate the effect of sex and dietary nitrate on COVID-19 vaccine-induced vascular dysfunction in healthy men and women: protocol of the DiNOVasc-COVID-19 study. Trials. 2023 Sep 16;24(1):593. doi: 10.1186/s13063-023-07616-2. PMID 37715222